CLINICAL TRIAL: NCT02265341
Title: Pilot Study of Ponatinib in Biliary Cancer Patients With FGFR2 Fusions
Brief Title: Ponatinib Hydrochloride in Treating Patients With Advanced Biliary Cancer With FGFR2 Fusions
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1345; NCI-2014-02075 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1345 (Other: Mayo Clinic in Arizona); P30CA015083 (NIH)
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2019-04

CONDITIONS: Malignant Hepatobiliary Neoplasm
MeSH Terms: interventions — ponatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (ponatinib hydrochloride) (Experimental): Patients receive ponatinib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Ponatinib Hydrochloride; Other: Quality-of-Life Assessment

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Ponatinib Hydrochloride — Given PO
  Other Names: AP24534 HCl
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This pilot phase II trial studies how well ponatinib hydrochloride works in treating patients with biliary cancer that has spread to other places in the body and that have alterations (fusions) in a gene known as fibroblast growth factor receptor 2 (FGFR2). Ponatinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the clinical benefit rate (confirmed complete or partial response or stable disease for 4 or more cycles) of ponatinib (ponatinib hydrochloride) in fibroblast growth factor receptor (FGFR) aberrant advanced biliary cancers.

SECONDARY OBJECTIVES:

I. To estimate progression free survival, overall survival, and cancer antigen 19-9 (CA19-9) response rate of these patients.

II. To estimate the adverse event profile of ponatinib.

TERTIARY OBJECTIVES:

I. Establish preliminary correlations between FGFR2 fusions and evidence of any clinical benefit.

II. Assess preliminary evaluation of FGFR2 pathway perturbation with ponatinib. III. To describe patient-reported health-related quality of life and symptoms.

OUTLINE:

Patients receive ponatinib hydrochloride orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for at least 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological confirmation of biliary cancer
* Confirmation of advanced biliary cancer that is refractory or intolerant to gemcitabine or fluoropyrimidine based therapy with FGFR2 fusion [using next-gen sequencing assays (such as Foundation One) or fluorescent in situ hybridization (FISH) break-apart assays] or FGFR pathway mutation/amplification [using next-gen sequencing assays (such as Foundation One)]; assays must be performed in a Clinical Laboratory Improvement Amendments [CLIA] certified laboratory and done as a CLIA validated test or research use only [RUO] in a CLIA laboratory
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Hemoglobin >= 9.0 g/dL
* Total bilirubin =< 1.5 x upper limit of normal (ULN), unless due to Gilbert's syndrome
* Aspartate transaminase (AST) and alanine aminotransferase (ALT) < 3 x ULN
* Creatinine =< 1.5 x ULN
* Serum lipase and amylase =< 2.5 x ULN; NOTE: if subject has tumor involvement in the liver =< 3 x ULN
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Recovered from prior radiotherapy and/or systemic therapy related toxicities to grade =< 1
* Provide informed written consent
* Life expectancy >= 3 months
* Willing to return to enrolling institution for follow-up (during the Active Monitoring Phase of the study); Note: during the Active Monitoring Phase of a study (i.e., active treatment and observation), participants must be willing to return to the consenting institution for follow-up
* Female and male patients who are fertile agree to use an effective form of contraception with their sexual partners from registration through 4 months after the end of treatment
* Ability to complete questionnaire(s) by themselves or with assistance

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients and patients known to be human immunodeficiency virus (HIV) positive and currently receiving antiretroviral therapy; NOTE: patients with a known history of HIV infection are not eligible for this trial
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Prior systemic chemotherapy, radiation therapy or major surgery =< 30 days prior to registration
* Concurrent use of any other approved or investigational anticancer agents, including hormonal agents
* Prior nitrosourea or mitomycin C =< 6 weeks prior to registration
* Patients with gastrointestinal comorbidities that would affect intake or absorption of ponatinib
* Untreated or progressive brain metastases
* Prior treatment with or allergic reactions attributed to compounds of similar chemical or biologic composition to ponatinib
* Clinically uncontrolled hypertension (diastolic blood pressure > 90 mm mercury [Hg]; systolic > 140 mm Hg); Note: patients with hypertension should be undergoing treatment at study entry for blood pressure control
* Previous or concurrent malignancy except adequately treated basal or squamous cell skin cancer, in situ carcinoma of the cervix, or other solid tumor treated curatively and without evidence of recurrence for at least 5 years
* History of significant bleeding disorder unrelated to cancer
* History of acute pancreatitis within 1 year prior to registration, chronic pancreatitis, alcohol abuse or uncontrolled hypertriglyceridemia (triglycerides > 450 mg/dL)
* Clinically significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

  * Any history of myocardial infarction, stroke, or revascularization
  * Unstable angina or transient ischemic attack within 6 months prior to registration
  * Congestive heart failure within 6 months prior to registration, or left ventricular ejection fraction (LVEF) less than lower limit of normal per local institutional standards within 6 months prior to registration
  * History of clinically significant (as determined by the treating physician) atrial arrhythmia
  * Any history of ventricular arrhythmia
  * Active venous thromboembolism including deep venous thrombosis or pulmonary embolism that is not amenable to treatment with anticoagulants
  * Patients with congenital prolonged QT syndromes and abnormal baseline prolonged corrected QT (QTc) (> 450 ms in men and > 470 ms in women)
  * Patients with an ejection fraction =< 50% as assessed by a baseline echocardiogram
* Taking medications that are known to be associated with torsades de pointes
* Taking any medications or herbal supplements that are known to be strong inhibitors of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) =< 14 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2019-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitesh Borad, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

REFERENCES:
- [Derived] Borad MJ, Gores GJ, Roberts LR. Fibroblast growth factor receptor 2 fusions as a target for treating cholangiocarcinoma. Curr Opin Gastroenterol. 2015 May;31(3):264-8. doi: 10.1097/MOG.0000000000000171. PMID 25763789
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ponatinib Hydrochloride)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ponatinib Hydrochloride)
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 48.5 [40.0 to 66.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 3
    1 | 7
    2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (Percentage), Which Includes Confirmed Tumor Response (Complete Response [CR] or Partial Response [PR]) or Stable Disease (SD)
Description: A confirmed tumor response is defined to be either a CR or PR noted as the objective status on 2 consecutive evaluations at least 8 weeks apart. The proportion of clinical benefit rate will be estimated by the number of patients with clinical benefit (confirmed CR, confirmed PR, or SD for 4 or more cycles) divided by the total number of evaluable patients. Complete Response (CR): All of the following must be true:a. Disappearance of all target lesions. b. Each target lymph node must have reduction in short axis to <1.0 cm. Partial Response (PR): At least a 30% decrease in PBSD (sum of the longest diameter for all target lesions plus the sum of the short axis of all the target lymph nodes at current evaluation) taking as reference the BSD (see Section 11.41). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for PD taking as reference the MSD. Please refer to RECIST v1.1 response criteria for more details.
Time Frame: Up to 10 months of treatment
Population: Only patients who received treatment for at least 8 weeks are evaluable for this outcome (i.e. one patient refused further treatment and was therefore unevaluable for response at 8 weeks)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Ponatinib Hydrochloride)
Number analyzed (Participants) | 11
percentage of patients | 45.5 [16.8 to 76.6]

2. Secondary Outcome: CA 19-9 Response
Description: This test measures the amount of a protein called CA 19-9 (cancer antigen 19-9) in the blood. CA 19-9 is a type of tumor marker. Tumor markers are substances made by cancer cells or by normal cells in response to cancer in the body.CA 19-9 was collected at baseline and on day one of each cycle. A CA 19-9 response is defined to be a >= 50% reduction from baseline. The CA 19-9 response rate (percentage) will be estimated by the number of CA 19-9 responses divided by the total number of evaluable patients.
Time Frame: Up to 10 months of treatment
Population: Only patients who had baseline and subsequent CA 19-9 levels measured in the study are evaluable for this analysis.
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Ponatinib Hydrochloride)
Number analyzed (Participants) | 3
percentage of patients | 0

3. Secondary Outcome: Overall Toxicity Rate, Assessed Using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0 (v4)
Description: The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns within patient groups. In addition, we will review all adverse event data that is graded as 3, 4, or 5 and classified as either "unrelated" or "unlikely to be related" to study treatment in the event of an actual relationship developing. The overall toxicity rates (percentages) for grade 3 or higher adverse events considered at least possibly related to treatment are reported below.
Time Frame: Up to 10 months of treatment
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Ponatinib Hydrochloride)
Number analyzed (Participants) | 12
percentage of patients | 41.7

4. Secondary Outcome: Progression-free Survival
Description: Progression free survival (PFS) is defined as the time from the date of registration to the date of disease progression or death resulting from any cause, whichever comes first. Progression is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Time from registration to the earliest date of documentation of disease progression, assessed up to maximum 3.3 years from registration.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ponatinib Hydrochloride)
Number analyzed (Participants) | 12
months | 2.4 [1.9 to 9.2]

5. Secondary Outcome: Survival Time
Description: Overall survival time is defined as the time from registration to death due to any cause. The median and 95% confidence intervals are estimated using the Kaplan-Meier estimator.
Time Frame: Time from registration to death due to any cause, assessed up to a maximum of 3.3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Ponatinib Hydrochloride)
Number analyzed (Participants) | 12
months | 15.7 [6.1 to NA] — The 95% Confidence interval upper limit was not able to be estimated due to an insufficient number of participants with events.

6. Other Pre Specified Outcome: Changes in Patient-reported Outcomes (Quality of Life and Symptoms), Assessed by the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30, EORTC QLQ-BIL21, Skindex-16, and Bowel Function Questionnaire
Description: The Uniscale assessment of overall quality of life will be used. The Was It Worth It questionnaire will determine patient's satisfaction with the study. Scale score trajectories over time will be examined using stream plots and mean plots with standard deviation error bars overall. Changes from baseline at each cycle will be statistically tested using paired t-tests, and standardized response means will be interpreted using Cohen's (1988) cut-offs. Correlation between outcomes will employ Pearson and/or Spearman correlations at individual time points.
Time Frame: Up to a maximum follow-up of 3.3 years
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Rate of Circulating-free Tumor Deoxyribonucleic Acid Mutations
Description: Will be described, and association with confirmed tumor response and/or clinical benefit will be investigated using a Fisher's exact test.
Time Frame: Up to a maximum follow-up of 3.3 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Rate of FGFR Fusions
Description: as for outcome 7
Time Frame: Up to a maximum follow-up of 3.3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to a maximum of 10 months on treatment.
Description: Each CTCAE term is a representation of a specific event used for medical documentation & analysis & is a single MedDRA Lowest Level Term (LLT). All graded AEs are reported for all patients. Serious AE (SAE) reports may include any secondary serious or non-serious events considered related to the primary event (the reason for filing an expedited report); collectively, these events are referred to as Expedited AEs, & appear in the SAE table.
Arm/Group | Treatment (Ponatinib Hydrochloride)
All-Cause Mortality (participants affected / at risk) | 9/12
Serious Adverse Events (participants affected / at risk) | 5/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ponatinib Hydrochloride) (N=12)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ponatinib Hydrochloride) (N=12)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 7 (17)
Constipation (Gastrointestinal disorders) | 7 (21)
Diarrhea (Gastrointestinal disorders) | 3 (7)
Nausea (Gastrointestinal disorders) | 6 (18)
Vomiting (Gastrointestinal disorders) | 2 (5)
Edema limbs (General disorders) | 5 (11)
Fatigue (General disorders) | 9 (41)
Fever (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3)
Alkaline phosphatase increased (Investigations) | 4 (8)
Blood bilirubin increased (Investigations) | 1 (2)
CD4 lymphocytes decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 5 (22)
White blood cell decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 7 (21)
Hypertension (Vascular disorders) | 3 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-04-13): https://cdn.clinicaltrials.gov/large-docs/41/NCT02265341/Prot_SAP_000.pdf